CLINICAL TRIAL: NCT02612389
Title: Meditative Movement for COPD Symptoms in Non-Smoking Flight Attendants
Acronym: MMforFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Flight Attendant Medical Research Institute (Other); ZRT Laboratory (Other); Norris Cotton Cancer Center (Other)
Responsible Party: Principal Investigator, Margaret A. Crane, Research Scientist, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28572
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Disease; Autonomic Dysfunction; COPD
Keywords: COPD; Qigong; ANS; Meditative Movement; Flight Attendants; Secondhand Smoke; Nicotine; Blood Pressure; 6 minute walk test
MeSH Terms: conditions — Lung Diseases; Primary Dysautonomias; Pulmonary Disease, Chronic Obstructive | interventions — Qigong

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MM Intervention taught via DVD (Experimental): Receive Meditative Movement training via DVD with pre and post interventional testing.
  Interventions: Other: Meditative Movement taught via DVD
- MM Intervention Waitlist Control (No Intervention): Testing at same frequency as Meditative Movement interventional subjects.

INTERVENTIONS:
Other: Meditative Movement taught via DVD — Gentle movement with attention to posture and breathing with emphasis on interoceptive awareness and self regulation.
  Other Names: Qigong
  Arms: MM Intervention taught via DVD

SUMMARY:
This study will explore the a Qigong based exercise intervention, here referred to as Meditative Movement (MM), to ameliorate the symptoms associated with chronic obstructive pulmonary disease (COPD) and its co-morbidities. It tests the hypothesis that MM will have a beneficial effect on COPD in FA, particularly on functional ability, respiratory symptoms, affective state, inflammation, and autonomic imbalance. If the hypothesis is correct, MM could be rapidly and inexpensively taught to FA with COPD and other COPD patients to slow degeneration and improve quality of life.

DETAILED DESCRIPTION:
The study has three phases.

Phase 1 will identify the best MM practices and their impact on a test group of affected FA. Phase 2 will develop a video to apply what is learned in Phase 1 to a larger group of affected FA, and will document the resulting impact on various aspects of pulmonary dysfunction and its comorbidities. Phase 3 is to refine the protocols and methods developed in earlier phases.

Phase 1: To identify the best set of MM exercises for improving COPD-related symptoms. This will be done by conducting a 12-week in-person MM program that will be held in one or more locations in the Northeastern region of the US and possibly other regions of the country.These training sessions will be used to determine precisely which MM exercises are most appropriate for this group. Selection will be based on professional judgment, participant feedback, and objective pre- and post-intervention measurements taken at the beginning and end of the 12-week program.

Phase 2: To use an RCT to evaluate the effectiveness of the exercises selected in Aim 1, as delivered by video only. We will design and produce an instructional DVD based on the findings in Aim 1.In the RCT we will test the hypothesis that targeted MM training and practice using the DVD alone will improve QOL, exercise tolerance, autonomic balance and pulmonary function, and reduce fatigue, in flight attendants with a COPD diagnosis. Pre- and post-intervention measurements will be compared, and to outcomes from a control group of flight attendants who will be wait listed for later participation in the study.

Phase 3: The videos used to train subjects in Phase II will be refined and the order of introduction of training modules will be adjusted. Efficacy will again be tested in newly recruited subjects. This is also a RCT.

ELIGIBILITY:
Inclusion Criteria:

* Occupation as a flight attendant for at least 5 years
* No history of significant tobacco use
* Occupational controls

Exclusion Criteria:

* Inability to give consent
* History of tobacco habituation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-03; Primary Completion 2020-06-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute walk test | Baseline, 4 months
  Each participant walks as many ft as possible at a brisk pace. The amount of feet covered in 6 minutes is documented.
Change in C-reactive protein (CRP) | Baseline, 4 months
  At each assessment circulating CRP will be monitored via blood collected in form of fingerstick.

SECONDARY OUTCOMES:
Blood Pressure | Baseline, 4 months
  Systolic and diastolic blood pressure, pre and post 6 minute walk test
Heart Rate | Baseline, 4 months
  Heart rate measured pre and post 6 minute walk test
Oxygen Saturation | Baseline, 4 months
  O2 saturation measured pre and post 6 minute walk test
Spirometry: FEV1/FVC | Baseline, 4 months
  Spirometric measurement of FEV1/FVC administered using EasyOne Spirometer. FEV1/FVC is the ratio of Forced Expiratory Volume (1sec)/FVC (Forced Vital Capacity, (Expiratory))
Autonomic Function Self Report | Baseline, 4 months
  Compass-31 administered via individual self-report.
Zung Anxiety Scale | Baseline, 4 months
  Zung anxiety questionnaire administered via individual self report.
Zung Depression Scale | Baseline, 4 months
  Zung depression questionnaire administered via individual self report.
Diurnal Salivary Cortisol | Baseline, 4 months
  4 sputum samples collected from subjects
Melatonin | Baseline, 4 months
  Melatonin levels from urine samples
Nicotine Exposure Autonomic Respiratory Syndrome (NEARS) | Baseline, 4 months
  New questionnaire under evaluation to reflect autonomic influences on respiratory and other physiologic functions in nicotine exposed study population. Range and meaning of range are yet to be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Steven N Fiering, PhD, Principal Investigator — Geisel School of Medicine, Faculty
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Zhang L, Xu Y. Impact of Radiation Therapy on Outcomes of Artificial Urinary Sphincter: A Systematic Review and Meta-Analysis. Front Surg. 2022 Feb 14;9:825239. doi: 10.3389/fsurg.2022.825239. eCollection 2022. PMID 35237650
- [Derived] Ye X, Gu Y, Bai Y, Xia S, Zhang Y, Lou Y, Zhu Y, Dai Y, Tsoi JK, Wang S. Does Low-Magnitude High-Frequency Vibration (LMHFV) Worth for Clinical Trial on Dental Implant? A Systematic Review and Meta-Analysis on Animal Studies. Front Bioeng Biotechnol. 2021 Apr 27;9:626892. doi: 10.3389/fbioe.2021.626892. eCollection 2021. PMID 33987172
- [Derived] Payne P, Fiering S, Zava D, Gould TJ, Brown A, Hage P, Gaudet C, Crane-Godreau M. Digital Delivery of Meditative Movement Training Improved Health of Cigarette-Smoke-Exposed Subjects. Front Public Health. 2018 Oct 19;6:282. doi: 10.3389/fpubh.2018.00282. eCollection 2018. PMID 30406067
- [Derived] Payne P, Fiering S, Leiter JC, Zava DT, Crane-Godreau MA. Effectiveness of a Novel Qigong Meditative Movement Practice for Impaired Health in Flight Attendants Exposed to Second-Hand Cigarette Smoke. Front Hum Neurosci. 2017 Feb 21;11:67. doi: 10.3389/fnhum.2017.00067. eCollection 2017. PMID 28270757
- [Derived] Payne P, Zava D, Fiering S, Crane-Godreau M. Meditative Movement as a Treatment for Pulmonary Dysfunction in Flight Attendants Exposed to Second-Hand Cigarette Smoke: Study Protocol for a Randomized Trial. Front Psychiatry. 2016 Mar 22;7:38. doi: 10.3389/fpsyt.2016.00038. eCollection 2016. PMID 27047398
- See also: Payne P, et al. (2016) Meditative Movement as a Treatment for Pulmonary Dysfunction in Flight Attendants Exposed to Second-Hand Cigarette Smoke: Study Protocol for a Randomized Trial. Front. Psychiatry 7:38. doi: 10.3389/fps — https://www.frontiersin.org/articles/10.3389/fpsyt.2016.00038/full
- See also: Payne P, et al. (2017) Effectiveness of a Novel Qigong Meditative Movement Practice for Impaired Health in Flight Attendants Exposed to Second-Hand Cigarette Smoke. Front. Hum. Neurosci. 11:67. doi: 10.3389/fnhu — https://www.frontiersin.org/articles/10.3389/fnhum.2017.00067/full
- See also: Payne P, Fiering S, Zava D, Gould TJ, Brown A, Hage P, Gaudet C and Crane-Godreau M (2018) Digital Delivery of Meditative Movement Training Improved Health of Cigarette-Smoke-Exposed Subjects. Front. Public Health 6:282. doi: 10.3389/fpubh.2018.00282 — https://www.frontiersin.org/articles/10.3389/fpubh.2018.00282/full
- See also: Website for Body Mind Science. Investigators are no longer at Dartmouth. Future publication links will be at the BodyMind Science sites. — http://www.bodymindscience.info